CLINICAL TRIAL: NCT04247425
Title: A Resistance Training Program to Improve Physical Function in Sarcoma Survivors
Brief Title: Progressive Resistance Training for the Improvement of Physical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lara Davis, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00019942; NCI-2019-05865 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-19103-L (Other: OHSU Knight Cancer Institute); STUDY00019942 (Other: OHSU Institutional Review Board); P30CA069533 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (resistance training, exercise counseling) (Experimental): Patients complete a series of progressive resistance training exercises at home twice weekly over 1 hour and receive instructional guidance from an exercise physiologist via videoconferencing once per week during one of these sessions for up to 12 weeks.
  Interventions: Other: Exercise Counseling; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Exercise Counseling — Receive instructional guidance
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Complete progressive resistance training
  Other Names: Strength Training

SUMMARY:
This trial studies how well progressive resistance training works in improving the physical function of sarcoma survivors. Treatments for sarcoma can cause side effects such as fatigue, muscle loss, and weakness, which can negatively impact a patient's ability to physically function and enjoy an independent lifestyle. Engaging in a resistance training exercise routine may improve physical function, body composition, and bone density of sarcoma survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of a home-based individualized progressive resistance training (PRT) program in sarcoma survivors.

SECONDARY OBJECTIVES:

I. To assess secondary measures of feasibility of a home-based, individualized PRT program in sarcoma survivors.

II. To determine if a 3-month PRT program improves physical function in sarcoma survivors.

EXPLORATORY OBJECTIVE:

I. To determine if a 3 month resistance training program improves body composition and bone mineral density.

OUTLINE:

Patients complete a series of progressive resistance training exercises at home twice weekly over 1 hour and receive instructional guidance from an exercise physiologist via videoconferencing once per week during one of these sessions for up to 12 weeks.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the Sarcoma Survivorship Registry (Institutional Review Board [IRB] #12039)

  * History of histologically-confirmed sarcoma
  * History of treatment with surgery, radiation and/or chemotherapy for the sarcoma diagnosis
  * Completion of sarcoma treatment >= 2 years prior to study enrollment
  * No evidence of recurrent or residual disease on surveillance exam or imaging for at least 2 years prior to study enrollment
* Sarcoma location must have been in the extremities, body wall, pelvic/shoulder girdle or axial skeleton. Intra-thoracic, intra-abdominal or cranial sarcomas are not eligible
* Currently engaging in < 1 hour of resistance exercise per week by self-report. Examples of resistance exercise include: using free weights or weight machines, push-ups, sit-ups, lunges, plank, etc.
* Able and willing to commit to attending weekly video coaching sessions and independently completing weekly resistance training sessions. This requires access to internet and a device with video and audio capabilities. A webcam may be provided by the study to the participant if needed
* Able and willing to commit to attending one initial in-person training session and one in-person follow-up assessment
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Medical contraindication(s) to any and all resistance training as determined by treating physician
* Non-English speaking. At this time, we do not have resources to support translation of exercise physiologist (EP) sessions
* Dependent on a mobility device (e.g., crutches, wheelchair) for independent activities of daily living (IADLs)

  * Use of a cane is permitted
* Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of participant safety or study results (e.g., pregnancy)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara E Davis, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Number of evaluable participants who completed end-of-intervention assessments
Time Frame: From the time of enrollment up to 3 months end-of-intervention assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
Participants | 9

2. Primary Outcome: Exercise Adherence
Description: Number of participants who completed end-of-intervention assessments and completed at least 18 of 24 prescribed training sessions.
Time Frame: From the time of enrollment up to completion of 12 week exercise intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 9
Participants | 7

3. Primary Outcome: Frequency of Related Serious Adverse Events (SAEs)
Description: Number of participants that experienced exercise-related SAEs
Time Frame: From the time of enrollment up to completion of 12 week exercise intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Individualized Progressive Resistance Training (PRT) Prescriptions
Description: Number of participants who received an individualized PRT prescription developed for the participant by the study exercise physiologist.
Time Frame: From the time of enrollment up to completion of 12 week exercise intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
Participants | 10

5. Secondary Outcome: Mean Patient-Reported Outcomes Measurement Information System (PROMIS) - Cancer Physical Function Score Value
Description: The PROMIS-Cancer assessment consists of 45 questions pertaining to physical function, each of which are designed as having five-point ordinal rating scales. Participants are asked to respond to questions regarding the extent of their physical function. Responses range from 1 to 5, where 1 represents "unable to do" and 5 represents "without any difficulty." Each PROMIS assessment generates a T-score, which is a standardized score with a mean of 50 and standard deviation of 10 in a reference population of cancer patients, i.e., a score of 40 is one SD lower than the mean of the reference population. A PROMIS-Cancer Physical Function score less than 50 indicates patient-reported physical function worse than the cancer patient mean. The PROMIS T-scores are summarized with mean and standard deviation, with comparison of scores at baseline and at 3 months using paired t-Test to determine if a 3-month resistance training program improves physical function.
Time Frame: Baseline up to completion of 12 week exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
score on a scale
  Baseline | 45.6 (9.4)
  End of Treatment | 47.2 (8.2)
Statistical Analysis 1: Comparison: Supportive Care (Resistance Training, Exercise Counseling); Baseline compared to end of 12 week exercise intervention; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Short Form-36 Physical Function Score
Description: The 36-Item Short Form Health Survey (SF-36) consists of a set of generic, quality-of-life measures to survey physical function in the general population. Responses range from 0 - 100, with a higher score indicating a more favorable health state. Will be summarized as mean and standard deviation. Will also compare scores at baseline and at 3 months using paired t-Test to determine if a 3-month resistance training program improves physical function.
Time Frame: Baseline up to completion of 12 week exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
score on a scale
  Baseline | 43.3 (8.4)
  End of Treatment | 49.1 (6.7)
Statistical Analysis 1: Comparison: Supportive Care (Resistance Training, Exercise Counseling); Baseline compared to end of 12 week exercise intervention; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Godin Leisure-Time Exercise Questionnaire Physical Activity Score (GLTEQ)
Description: To score the GLTEQ, the weekly frequencies of strenuous, moderate, and light activities are multiplied by nine, five, and three, respectively. Total weekly leisure activity is calculated in arbitrary units by summing the products of the separate components as shown in the following formula: Weekly leisure activity score = (9xStrenuous) + (5x Moderate) + (3xLight). Responses range from 0 - greater than 24, with 0 indicating no activity and a higher score indicating more activities (no maximum score). GLTEQ will be summarized as mean and standard deviation. Will also compare scores at baseline and at 3 months using paired t-Test to determine if a 3-month resistance training program improves physical function.
Time Frame: Baseline up to completion of 12 week exercise intervention
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
arbitrary units
  Baseline | 28.6 (32.9)
  End of Treatment | 20.8 (12.1)
Statistical Analysis 1: Comparison: Supportive Care (Resistance Training, Exercise Counseling); Baseline compared to end of 12 week exercise intervention; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy-Fatigue Score (FACT-F)
Description: Fatigue was assessed using the FACT-F scale. This is a 13 item, uni-dimensional, 5-point Likert scale, measuring physical fatigue over the past week. The scale has high internal consistency and is widely used in the literature. Responses range from 0 - 52, with a higher score indicating more fatigue. FACT-F will be summarized as mean and standard deviation. Will also compare scores at baseline and at 3 months using paired t-Test to determine if a 3-month resistance training program improves physical function.
Time Frame: Baseline up to completion of 12 week exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 10
score on a scale
  Baseline | 30.2 (14.8)
  End of Treatment | 40.1 (10)
Statistical Analysis 1: Comparison: Supportive Care (Resistance Training, Exercise Counseling); Baseline compared to end of 12 week exercise intervention; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Difference in 1-repetition Maximum (Kilogram)
Description: Compare scores at baseline and at 3 months using paired t-Test to determine if a 3-month resistance training program improves physical function. Will initially examine distribution of each outcome variable using Shapiro-Wilk test, as well as data visualization techniques as standard practice. Will consider transforming the data or adopting non-parametric approaches if normality assumption is violated.
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Short Physical Performance Battery Score
Description: as for outcome 9
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Grip Strength (Kilogram)
Description: as for outcome 9
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Gait and Balance
Description: Measured by mobile sensor. Will compare scores at baseline and at 3 months using paired t-Test to determine if a 3-month resistance training program improves physical function. Will initially examine distribution of each outcome variable using Shapiro-Wilk test, as well as data visualization techniques as standard practice. Will consider transforming the data or adopting non-parametric approaches if normality assumption is violated
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Instrumented 6-minute Walk Test
Description: as for outcome 9
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Instrumented Postural Sway
Description: as for outcome 9
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Instrumented Timed up and go Test
Description: as for outcome 9
Time Frame: Baseline up to completion of 12 week exercise intervention
Population: Data could not be collected due to COVID restrictions
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of consent until the end of treatment visit (12 weeks). Any clinically significant adverse events persisting at the end of treatment visit were followed until resolution, stabilization, or death, whichever came first.
Arm/Group | Supportive Care (Resistance Training, Exercise Counseling)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The COVID pandemic resulted in extensive protocol revisions to pivot from in person assessments to telehealth. Multiple secondary endpoints were therefore not collected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT04247425/Prot_SAP_ICF_000.pdf